CLINICAL TRIAL: NCT05298267
Title: Reducing Distracted Driving With the Flip of a Switch
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn prior to study launch because a research partnership with the school district could not be secured in time
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 851002
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Automobile Accident
Keywords: distracted driving automobile; behavioral economics (nudge); smartphone application

STUDY DESIGN:
Intervention Model Description: Participants will be monitored for 4 weeks. Halfway through the monitoring period, participants will be asked to turn on the DNDWD feature on their phone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring phase (Experimental): Participants will be monitored for 4 weeks. Halfway through the monitoring period, participants will be asked to turn on DNDWD.
  Interventions: Device: Do Not Disturb While Driving

INTERVENTIONS:
Device: Do Not Disturb While Driving — Participants will be asked to turn on Do Not Disturb While Driving on their smartphones.

SUMMARY:
We propose to test a potential intervention to reduce distracted driving among high school students that could be used as part of future research trials and school campaigns. This intervention is designed to encourage use of a setting that silences incoming calls and messages while the person is driving.

DETAILED DESCRIPTION:
The purpose of this study is to test an intervention to reduce distracted driving among high school students. We're interested in learning the use of Do Not Disturb While Driving (DNDWD) by high school students. Participants will be recruited to participate into a 4-week study. Those that consent will download a driving app that will monitor their phone use while driving. Halfway through the monitoring period, we will ask participants to turn on DNDWD. Participants will also have the opportunity to enroll into an auto-reply message contest for best message. Once the 4- week monitoring period is complete participants will complete and exit survey

ELIGIBILITY:
Inclusion Criteria:

1. High School student with school assigned email address
2. Has a cell phone with ability to download Way to Drive app
3. Has a driver's license and typically drives every week

Exclusion Criteria:

1. Unable to read or understand English
2. Under 18 years old and no parental consent

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported DNDWD | For the duration of the study; 4 weeks
  Change is reported use. Dichotomy of use or non-use pre and post intervention

SECONDARY OUTCOMES:
Seconds of active (handheld) phone use per hour of driving | For the duration of the study; 4 weeks
  This is a composite outcome that measures the proportion of total trip time in which the driver is engaged in handheld phone call use or non-call handheld use (e.g. texting, swiping, and typing), as measured by the Way to Drive app. Several studies (e.g. Klauer, NEJM, 2014) have demonstrated the association between handheld phone use (e.g., reaching for phone, typing, swiping, dialing) and increased crash risk. This outcome is also known as the active phone use percentage. Passive phone use (e.g. phone is streaming GPS navigation directions or music without any typing, swiping, and handheld holding of the phone) is not included in this outcome. Trips are only counted if the app predicts the user was a driver for the trip based on the phone sensor data and the user does not correct the app; or, if the user corrects the app and indicates they were driving.
Seconds of active (handheld) call use per hour of driving. | For the duration of the study; 4 weeks
  We will analyze the components of the secondary outcome separately.
Seconds of active (handheld) non-call use per hour of driving | For the duration of the study; 4 weeks
  We will analyze the components of the secondary outcome separately.
Seconds of passive (hands-free) call use per hour of driving | For the duration of the study; 4 weeks
  Use of DNDWD should also cut down on hands-free driving distraction.
Seconds of passive (hands-free) non-call use per hour of driving. | For the duration of the study; 4 weeks
  Use of DNDWD should also cut down on hands-free driving distraction.
Seconds of speeding per hour of driving | For the duration of the study; 4 weeks
  . Speeding events, defined as >10 mph above the posted speed limit, are detected by the app.
Hard braking events per 100 miles. | For the duration of the study; 4 weeks
  Hard braking events are detected by the app.
Fast acceleration events per 100 miles. | For the duration of the study; 4 weeks
  Fast acceleration events are detected by the app.
  Acceptability of interventions will be measured using a mixed-methods approach:
Net promoter score | For the duration of the study; 4 weeks
  In the exit survey, participants will be asked "How likely is it that you would recommend this program to a friend or colleague?" on a 0 to 10 scale.
Responses to open-ended questions in exit survey | For the duration of the study; 4 weeks
  Participants will be asked the following two open-ended questions: 1) "Please tell us what you liked about participating in this study;" 2) "Please tell us what you didn't like about participating in this study and how we should improve the experience in the future." These qualitative responses will be coded for content related to intervention acceptability and emerging themes will be identified.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asch DA, Rosin R. Engineering Social Incentives for Health. N Engl J Med. 2016 Dec 29;375(26):2511-3. doi: 10.1056/NEJMp1603978. No abstract available. PMID 28029924
- [Background] AT&T. AT&T Teen Driver Survey: Executive Summary 2012. https://www.att.com/Common/aboutus/txtingdriving/attteensurveyexecutive.pdf
- [Background] Delgado MK, Wanner KJ, McDonald C. Adolescent Cellphone Use While Driving: An Overview of the Literature and Promising Future Directions for Prevention. Media Commun. 2016 Jun 16;4(3):79-89. doi: 10.17645/mac.v4i3.536. PMID 27695663
- [Background] Department of Transportation, NHTSA. Visual-Manual NHTSA Driver Distraction Guidelines for Portable and Aftermarket Devices. 2016. Docket No. NHTSA-2013-0137. Available at: https://www.nhtsa.gov/press-releases/us-dot-proposes-guidelines- address-driver-distraction-caused-mobile-devices-vehicles.
- [Background] Creaser JI, Edwards CJ, Morris NL, Donath M. Are cellular phone blocking applications effective for novice teen drivers? J Safety Res. 2015 Sep;54:75-8. doi: 10.1016/j.jsr.2015.06.014. Epub 2015 Jul 29. PMID 26403905
- [Background] Ebel B, Boyle L, O'Connor S, et al. Randomized Trial of Cell Phone Blocking and In-Vehicle Camera To Reduce High-Risk Driving Events among Novice Drivers. San Diego, CA: Pediatric Academic Societies; 2015.
- [Background] Funkhouser D, Sayer JR. Cellphone Filter/Blocker Techonology Field Test. Washington, DC: NHTSA; 2013. Report No. HS 811 863.
- [Background] Hayashi Y, Russo CT, Wirth O. Texting while driving as impulsive choice: A behavioral economic analysis. Accid Anal Prev. 2015 Oct;83:182-9. doi: 10.1016/j.aap.2015.07.025. Epub 2015 Aug 13. PMID 26280804
- [Background] Holm S. A simple sequentially rejective multiple test procedure. Scandinavian J. of Statistics 1979 6:65-70.
- [Background] Kervick AA, Hogan MJ, O'Hora D, Sarma KM. Testing a structural model of young driver willingness to uptake Smartphone Driver Support Systems. Accid Anal Prev. 2015 Oct;83:171-81. doi: 10.1016/j.aap.2015.07.023. Epub 2015 Aug 13. PMID 26277411
- [Background] Kolko, Jed. "How Suburban Are Big American Cities?" FiveThirtyEight, 15 May 2015, fivethirtyeight.com/features/how-suburban-are-big-american-cities/.
- [Background] Klauer SG, Guo F, Simons-Morton BG, Ouimet MC, Lee SE, Dingus TA. Distracted driving and risk of road crashes among novice and experienced drivers. N Engl J Med. 2014 Jan 2;370(1):54-9. doi: 10.1056/NEJMsa1204142. PMID 24382065
- [Background] Loewenstein G, Asch DA, Volpp KG. Behavioral economics holds potential to deliver better results for patients, insurers, and employers. Health Aff (Millwood). 2013 Jul;32(7):1244-50. doi: 10.1377/hlthaff.2012.1163. PMID 23836740
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Musicant O, Lotan T. Can novice drivers be motivated to use a smartphone based app that monitors their behavior? Transp Res Part F Traffic Psy- chol Behav. 2016;42:544-557.
- [Background] National Highway Traffic Safety Administration. Distracted Driving 2014. Traffic Safety Facts Research Note. Available at: http://www.-nrd.nhtsa.dot.gov/CATS/index.aspx
- [Background] Richtel M. Phone makers could cut off drivers. So why don't they? New York Times. September 24, 2016.
- [Background] Sinder M. iPhone will get "Do Not Disturb While Driving" mode in iOS 11 this fall. USA Today. June 5, 2017.
- [Background] Using Technology to Fix the Texting-While-Driving Problem. National Public Radio. April 24, 2014.